CLINICAL TRIAL: NCT02024308
Title: A Randomized Comparison of Fludarabine in Combination With Cytarabine Versus High -Dose Cytarabine in Post-remission Therapy for AML1-ETO Acute Myeloid Leukemia
Brief Title: AML1-ETO Acute Myeloid Leukemia With Fludarabine and Cytarabine Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xianmin Song, Associate Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHXY-AML01
Record Dates: First submitted 2013-12-20; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Acute Myeloid Leukemia; AML1-ETO Fusion Protein Expression
Keywords: acute myeloid leukemia,; AML1-ETO fusion protein,; Fludarabine,; recurrence
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — fludarabine; fludarabine phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine (Experimental): The patients in experimental arm should receive the consolidation chemotherapy regimen with fludarabine and cytarabine. The dosage of fludarabine is 30mg/m2/d for 5 days intravenously and cytarabine is 1.4g/m2/d for 5 days intravenously.
  Interventions: Drug: Fludarabine; Drug: Cytarabine
- HD-Arac (Active Comparator): The patients in control arm should receive the consolidation chemotherapy regimen with high-dose cytarabine. The dosage of cytarabine is 2000mg/m2/12h for 3 days (1,3,5) intravenously.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Fludarabine — 50 mg/m2, IV (in the vein) in combination with cytarabine 1.4mg/m2/d for 5 days with each cycle of 28 days. Number of cycles: 4
  Other Names: Fludara
  Arms: Fludarabine
Drug: Cytarabine — 2000mg/m2/12h, IV (in the vein) for 3 days with each cycle of 28 days. Number of cycles: 4
  Other Names: Cytosar

SUMMARY:
The purpose of the study is to determine whether Fludarabine in combination with cytarabine is more effective than high-dose cytarabine in post-remission therapy for patients with AML1-ETO acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of AML1-ETO positive acute myeloid leukemia
* In status of complete remission after one to two courses of induction therapy with DA(Daunorubicin 60mg/m2/d for 3 days, cytarabine 100mg/m2/d for 5-7days) regimen
* ECOG (Eastern Cooperative Oncology Group) score: <2

Exclusion Criteria:

* Serious liver/ kidney dysfunction
* Cardiac function level: 2 above
* Female in pregnancy or lactation
* With serious infection diseases or other diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with disease recurrence | one year

SECONDARY OUTCOMES:
Percentage of Participants in survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, Doctor, Principal Investigator — Department of Hematology, Changhai Hospital
Locations (1):
- Department of Hematology, Changhai Hospital, Shanghai, China